CLINICAL TRIAL: NCT04198623
Title: A Phase II Study, Evaluating the Efficacy of Montelukast in Reducing the Incidence and Severity of Monoclonal Antibodies Associated Infusion Reactions
Brief Title: Efficacy of Montelukast in Reducing the Incidence and Severity of Monoclonal Antibodies Associated Infusion Reactions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mohammed Bukari, MD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2019105; IND146287 (Other: US FDA)
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Infusion Reaction; Monoclonal Antibody
MeSH Terms: interventions — montelukast; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Montelukast (Singulair) (Other): Montelukast(Singulair) 10mg to be taken in addition to standard institutional premedication
  Interventions: Drug: Montelukast 10 Mg Oral Tablet

INTERVENTIONS:
Drug: Montelukast 10 Mg Oral Tablet — Montelukast(Singulair) 10mg to be taken at least 2 hours prior to initiation of monoclonal antibody infusion addition to institutional protocol premedication regiment
  Other Names: Singulair

SUMMARY:
The use of monoclonal antibodies (MA) either alone or as part of chemoimmunotherapy in oncology, benign and malignant hematology is expanding. Of the 17 therapeutic MAs approved in 2017 by FDA, 50% of them are indicated for hematologic and oncologic condition. With increasing number of approved agents, therapeutic MAs have become one of the fastest growing areas in the management of benign and malignant hematologic condition. Advancement of recombinant technology allows development of partially or fully humanized new agents. Despite this, they still carry significant risk of immune and non-immune mediated adverse events. Most of the therapeutic monoclonal antibody related adverse events (MCAAE) The severity of reaction is variable, ranging from mild involvement of single organ to severe and life-threatening reactions requiring hospitalization or even resulting in death.

Even for mild infusion reactions, where re-initiation of infusion is possible, there is resultant delay in delivery of infusions, distress to patients, and additional utilization of health care resources.

Due to unpredictability of standard infusion reaction (SIR), efforts have been focused on premedication to decreasing the incidence and severity of infusion reaction. Most institutions have protocols using corticosteroid, acetaminophen and antihistamine as part of their premedication protocols. This has reduced but not eliminated standard infusion reactions. Most recently, mast cell stabilizers are being added to standard protocols to further reduce the incidence and severity of standard infusion reactions with variable anecdotal success without formal study. Of all the monoclonal antibodies, only Daratumumab has been evaluated using this strategy.

This study seeks to evaluate the efficacy of mast cell stabilizer Montelukast (SINGULAIR) 10 mg in decreasing the SIR in patients receiving therapeutic MAs either alone or as part of chemoimmunotherapy in hematologic condition. The MAs being studied includes: Blinatumomab (BLINCYTO, Amgen Inc.), Daratumumab (DARZALEX, Janssen Biotech, Inc.), Elotuzumab (EMPLICIT, Bristol-Myers Squibb Company), Gemtuzumab (MYLOTARG, Pfizer Inc.), Obinutuzumab (GAZYVA, Genentech USA, Inc.), and Rituximab (RITUXAN, Genentech US); The investigators postulate that 10 mg of Montelukast, when given in addition to standard premedication, will lead to decrease in incidence of MA associated SIR, shorter infusion time and decrease use of additional health care resources

DETAILED DESCRIPTION:
Study design:

This is a Phase II single arm open label study evaluating 10 mg Montelukast given at least 2 hours prior to infusion of monoclonal antibody in addition to standard premedication. Monoclonal antibodies being evaluated include those commonly used to treat hematologic and oncologic malignancies like (Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab).

Arms/Intervention; Study subjects will be given 10 mg of Montelukast to be orally self-administered at least 2 hours prior to beginning of chemotherapy section Standard premedication will be administered according to institution protocol

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years.
2. Able to provide consent for study participation (English and Spanish).
3. Patients with hematologic disorders or malignancies starting on any of the following monoclonal antibodies alone or in combination with chemotherapy (Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab).
4. Able to tolerate leukotriene antagonist including Montelukast.
5. Able to tolerate oral intake.
6. Available for follow up by phone and on site.

Exclusion Criteria:

1. Patients undergoing treatment with above monoclonal antibodies for indications other than stated in above eligibility criteria.
2. Patients who cannot provide informed consent in English or Spanish.
3. Patients taking Montelukast or other leukotriene antagonists for other indications at the time of screening.
4. Known allergic reactions to Montelukast or other leukotriene inhibitors.
5. On monoclonal antibodies other than the ones being studied (Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab).
6. History of uncontrolled depression or suicidal ideation or psychiatric illness.
7. Known Severe Hepatic Impairment (AST>10x ULN; ALT>10x ULN; ALP>10x ULN; and/or Bilirubin >5x ULN).
8. Patient with eosinophilic vasculitis.
9. Unable to comply with phone or in person follow-up.
10. Patients participating in another clinical trial.
11. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMMED BUKARI, MD, Principal Investigator — UCSF - Fresno
Locations (1):
- Community Cancer Institute, Clovis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Incidence rate of Infusion reaction Tolerability of infusion reaction
Supporting Information: CSR
Time Frame: Sept, 2022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hematology and Oncology Clinic of Community Cancer Institute
Pre-assignment Details: Patients with hematologic disorders or malignancies starting on any of the following monoclonal antibodies alone or in combination with chemotherapy (Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab
Groups:
- Open Label Single Arm Treatment Group: Phase II single arm open label study evaluating 10 mg Montelukast given at least 1 hour prior to infusion of each dose of Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab) in addition to standard premedication up to 6 doses
Period: Overall Study
Arm/Group | Open Label Single Arm Treatment Group
Started | 40
Completed | 39
Not Completed | 1
Not completed — 1 patient was taken off due to covid-19 pandemic shut down | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Single Arm Treatment Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Medication allergy [Count of Participants; unit: Participants]
  At least 1 medication allergy | 15
  No Medication allergy | 25
At least 1 Atopic Condition ( [Count of Participants; unit: Participants]
  Present | 7
  Absent | 33
Monoclonal Antibody Treatment [Count of Participants; unit: Participants]
  Rituximab | 21
  Daratumumab | 7
  Blinatumomab | 3
  Gemtuzumab | 5
  Elotuzumab | 1
  Obinutuzumab | 3
Diagnosis [Count of Participants; unit: Participants]
  Follicular lymphoma | 3
  Diffuse Large B cell Lymphoma | 12
  Marginal Zone Lymphoma | 4
  Multiple Myeloma/amyloidosis | 8
  CLL | 2
  ALL | 3
  AML | 6
  ITP/AIHA | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Standard Infusion Reactions (SIR) at Cycle 1 and During Subsequent Cycles of Monoclonal Antibody Infusion
Description: The incidence rate of infusion reaction includes all clinical sign and symptoms of reaction graded by CTCAE v5.0 in patients receiving each cycle monoclonal antibody infusions. The grade and rate of each grade will be measured and or calculated for each cycle of infusion up to 6 cycles or treatment discontinuation which ever comes first
Time Frame: Through study completion (average 6 months)
Population: The incidence rate of all grades of infusion reaction on the day of infusion during or after administration of cycle 1 of Monoclonal Antibody treatment in all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast (Singulair)
Number analyzed (Participants) | 40
Participants
  Cycle 1 infusion reaction: Infusion reaction | 14
  Cycle 1 infusion reaction: No infusion reaction | 26
  Cycle 2-6 infusion reaction: number analyzed (Participants) | 39
  Cycle 2-6 infusion reaction: Infusion reaction | 4
  Cycle 2-6 infusion reaction: No infusion reaction | 35

2. Secondary Outcome: Average Infusion Duration of Each Cycle of the Monoclonal Antibody Infusion in the Study Subject
Description: The time from start to end of each cycle of infusion of monoclonal antibody will be measured in the study subject up to 6 cycles or treatment discontinuation which ever comes first. Average infusion time will then be calculated.
Time Frame: Through study completion (average 6 months)
Population: Total population is separated to the differing monoclonal antibody treatment regimen
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Number of infusion
Groups:
- Open Label Single Arm Treatment Group - Cycle 1 Infusion; Open Label Single Arm Treatment Group - Cycles 2-6: Phase II single arm open label study evaluating 10 mg Montelukast given at least 1 hour prior to infusion of each dose of Blinatumomab, Daratumumab, Elotuzumab, Gemtuzumab, Obinutuzumab, and Rituximab) in addition to standard premedication up to 6 doses
Arm/Group | Open Label Single Arm Treatment Group - Cycle 1 Infusion | Open Label Single Arm Treatment Group - Cycles 2-6
Number analyzed (Participants) | 40 | 40
Number analyzed (Number of infusion) | 40 | 152
minutes
  Rituximab infusions: number analyzed (Participants) | 21 | 21
  Rituximab infusions: number analyzed (Number of infusion) | 21 | 76
  Rituximab infusions | 267.0 (151.0) | 194.0 (70.3)
  Obinutuzumab infusions: number analyzed (Participants) | 3 | 3
  Obinutuzumab infusions: number analyzed (Number of infusion) | 3 | 15
  Obinutuzumab infusions | 311.0 (56.0) | 218.5 (18.0)
  Daratumumab infusions: number analyzed (Participants) | 7 | 7
  Daratumumab infusions: number analyzed (Number of infusion) | 7 | 33
  Daratumumab infusions | 110.0 (132.0) | 87.4 (103.7)
  Gemtuzumab infusions: number analyzed (Participants) | 5 | 5
  Gemtuzumab infusions: number analyzed (Number of infusion) | 5 | 8
  Gemtuzumab infusions | 162.8 (59.7) | 292.4 (391.4)
  Blinatumomab infusions: number analyzed (Participants) | 3 | 3
  Blinatumomab infusions: number analyzed (Number of infusion) | 3 | 15
  Blinatumomab infusions | 60.0 (84.3) | 115.5 (244.0)
  Elotuzumab infusions: number analyzed (Participants) | 1 | 1
  Elotuzumab infusions: number analyzed (Number of infusion) | 1 | 5
  Elotuzumab infusions | 176 (NA) — Only one data point captured for this instance | 68.0 (11.4)

3. Secondary Outcome: Incidence Rate of Grade 3 or More Monoclonal Antibody Infusion Throughout the Entire Duration of Infusion (up to 6 Cycles or Till Discontinuation Whichever Comes First)
Description: The incidence rate of Grade 3 infusion reaction includes all clinical sign and symptoms of reaction graded by CTCAE v5.0 as grade 3 in patients receiving all monoclonal antibodies through out the entire duration of treatment(up to 6 cycles or till treatment is discontinue which ever comes first
Time Frame: Through study completion (average 6 months)
Population: Patient who had infusion reaction
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast (Singulair)
Number analyzed (Participants) | 40
Participants
  Infusion reactions (all grades) of cycle 1: Infusion reactions | 14
  Infusion reactions (all grades) of cycle 1: No infusion reactions | 26
  Infusion reactions (grade 3 or greater) of cycle 1: Infusion reactions | 4
  Infusion reactions (grade 3 or greater) of cycle 1: No infusion reactions | 36
  Infusion reactions (all grades) of cycle 2-6: Infusion reactions | 4
  Infusion reactions (all grades) of cycle 2-6: No infusion reactions | 36
  Infusion reactions (grade 3 or greater) of cycle 2-6: Infusion reactions | 0
  Infusion reactions (grade 3 or greater) of cycle 2-6: No infusion reactions | 40

4. Secondary Outcome: Discontinuation Rate of Monoclonal Antibody Infusion Due to SIRs
Description: Rate at which monoclonal antibody treatment is stopped and changed to new treatment due to adverse drug reaction attributed to monoclonal antibody infusion
Time Frame: Through study completion (average 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm Treatment Group
Number analyzed (Participants) | 40
Participants
  No | 37
  Yes | 3

5. Other Pre Specified Outcome: Infusion Data Cycle 1
Time Frame: Cycle 1
Measure: Count of Participants; unit: Participants
Groups:
- Open Label Single Arm Treatment Group: Breakdown of infusion drugs
Arm/Group | Open Label Single Arm Treatment Group
Number analyzed (Participants) | 40
Participants
  Rituximab | 21
  Daratumumab | 7
  Gemtuzumab | 5
  Obinutuzumab | 3
  Blinatumomab | 3
  Elotuzumab | 1

6. Other Pre Specified Outcome: Infusion Data Cycle 2-6
Time Frame: Cycle 2-6
Population: 1 patient was taken off study due to covid-19 pandemic and suspension of non-essential clinical trial
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm Treatment Group
Number analyzed (Participants) | 40
Participants
  Rituximab | 20
  Daratumumab | 7
  Gemtuzumab | 5
  Obinutuzumab | 3
  Blinatumomab | 3
  Elotuzumab | 1
  Removed from study | 1

ADVERSE EVENTS:
Time Frame: 6 months post start of cycle 1 of infusion
Description: National Cancer Institute Common Terminology of Standard Adverse Effect (NCI CTCAE v5.0)
Arm/Group | Montelukast (Singulair)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 12/40
Other Adverse Events (participants affected / at risk) | 2/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (Singulair) (N=40)
Infusion reaction (Immune system disorders) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (Singulair) (N=40)
National Cancer Institute Common Terminology of Standard Adverse Effect (NCI CTCAE v5.0) (Immune system disorders) | 2 (2) — Diarrhea, rash, nausea and vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04198623/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04198623/ICF_002.pdf